CLINICAL TRIAL: NCT02705469
Title: A Phase 1 Safety and Tolerability Study of ZEN003694 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of ZEN003694 in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zenith Epigenetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZEN003694-001
Record Dates: First submitted 2016-02-10; First posted 2016-03-10 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Metastatic Castration-Resistant Prostate Cancer
Keywords: Metastatic Castration-Resistant Prostate Cancer (mCRPC); Phase 1; Prostate Cancer; Pharmacokinetics (PK); ZEN003694; ZEN-3694; Metastatic Castrate-Resistant Prostate Cancer; BET inhibitor (BETi); Bromodomain; Pharmacodynamics (PD); Epigenetics
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Escalation and Dose Confirmation - ZEN003694 Single Agent (Experimental): ZEN003694 will be administered orally as a single agent once daily in 28-day cycles, enrolling mCRPC patients.
  Interventions: Drug: ZEN003694

INTERVENTIONS:
Drug: ZEN003694

SUMMARY:
This is an open label, Phase 1, dose escalation and dose confirmation study of ZEN003694 in patients with mCRPC.

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 years
2. Metastatic, castrate resistant, histologically confirmed prostate cancer; surgically castrated or continuous medical castration for ≥ 8 weeks prior to screening
3. Serum testosterone < 50 ng/dL determined within 4 weeks of first administration of study drug
4. Prior progression on one or more androgen-receptor/androgen-synthesis inhibitor therapies (e.g. abiraterone, enzalutamide, apalutamide, TAK-700 and/or galeterone) by Prostate Cancer Working Group 2 (PCWG2) criteria. Prior progression on bicalutamide/nilutamide/flutamide/ketoconazole alone is not allowed.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Adequate laboratory parameters [absolute neutrophil (ANC), platelets, aspartate aminotransferase (AST), alanine aminotransferase (ALT), total bilirubin, creatinine and coagulation parameters] at screening

Exclusion Criteria:

1. Any history of brain metastases or prior seizure or conditions predisposing to seizure activity
2. Have previously received an investigational BET inhibitor (including previous participation in this study or Study ZEN003694-002)
3. Have received prior systemic anti-cancer therapy or investigational therapy within 2 weeks or five half-lives, whichever is shorter, prior to the first administration of study drug
4. Failure to recover to Grade 1 or lower toxicity related to prior systemic therapy (excluding alopecia and neuropathy) prior to study entry
5. Radiation therapy within 2 weeks of first administration of study drug
6. Have received prior chemotherapy in the metastatic castration-resistant setting (prior chemotherapy in the hormone-sensitive setting is allowed provided last dose was at least 6 months prior to study entry)
7. Currently receiving medications known to be strong inducers or inhibitors of CYP3A4 with a narrow therapeutic window. Strong inducers and inhibitors of CYP3A4 with narrow therapeutic ranges must be discontinued at least 7 days prior to the first administration of study drug.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
For dose escalation only: Incidence of dose-limiting toxicities (DLT) | Cycle 1 (Day 1 thru Day 28)
  A DLT is a treatment-related, clinically significant adverse event or laboratory abnormality occurring during the first cycle of treatment (Day 1 thru Day 28).
For dose escalation and dose confirmation: Incidence of treatment-related adverse events (AE) and treatment-related serious adverse events (SAE) | Up to 24 months

SECONDARY OUTCOMES:
Measure the pharmacokinetic (PK) parameter: AUC of ZEN003694 | Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 2 Day 1: pre-dose
  AUC is defined as the area under the curve (plasma concentration of drug over time).
Measure the PK parameter: Cmax of ZEN003694 | Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 2 Day 1: pre-dose
  Cmax is defined as maximum or peak plasma concentration of drug.
Measure the PK parameter: Cmin of ZEN003694 | Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 2 Day 1: pre-dose
  Cmin is defined as minimum or trough plasma concentration of drug.
Measure the PK parameter: Tmax of ZEN003694 | Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 2 Day 1: pre-dose
  Tmax is defined as the time from dosing to the maximum plasma concentration.
Measure the PK parameter: t1/2 of ZEN003694 | Cycle 1 Day 1: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 1 Day 2: pre-dose; Cycle 1 Day 15: pre-dose, 0.25, 0.5, 1, 2, 4, 6 and 8 hours post-dose; Cycle 2 Day 1: pre-dose
  t/12 is defined as the half-life of drug.
Evaluate prostate-specific antigen (PSA) response rate by PCWG2 criteria | From screening up to 24 months
Evaluate radiographic response rate by PCWG2 criteria | From screening up to 24 months
Evaluate median progression-free survival by PCWG2 criteria | From screening up to 24 months
Evaluate circulating tumor cell (CTC) response rate during dose confirmation phase only | From screening up to 12 months

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California Los Angeles Medical Center, Los Angeles, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Karmanos Cancer Institute, Detroit, Michigan
  - Karmanos Cancer Institute, Farmington Hills, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Virginia Oncology Associates, Hampton, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No